CLINICAL TRIAL: NCT06913439
Title: Fin Wax Bath Therapy in Patients With Post-traumatic Stiffness of Knee Joint: A Randomized Controlled Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/799
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Stiffness; Sacroiliac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Active Comparator)
  Interventions: Diagnostic Test: Exercise Group
- Parafin Wax Bath (Experimental)
  Interventions: Combination Product: Parafin Wax Bath

INTERVENTIONS:
Diagnostic Test: Exercise Group — technique was implemented with three sets of ten repetitions on each treatment occasion for a period of 3 days/ week for 8 weeks. In this group, the adjustable couch was used to treat the patients effectively. During MWM, position of the patients was prone lying and high sitting position with swinging bilateral leg out of the couch at available various range of motion of affected knee joint. In prone lying position, the therapist was stand just behind the patient towards the affected knee joint. The mulligan belt placed at proximal tibia ends which already wrapped with the lower back of the therapist. In high or couch sitting position, the therapist was sitting on rest chair. The method using of mulligan belt was same as in prone lying position. After stabilization, the mobilization with movement (MWM) started in order with the therapist mobilized the knee joint followed by active movement of knee joint performed by the patients
  Arms: Exercise Group
Combination Product: Parafin Wax Bath — Group B will receive Paraffin Wax Bath Therapy in combination with standard care exercises. In this treatment, the affected knee joint will be immersed in warm paraffin wax to deliver thermotherapy, which helps reduce joint stiffness, improve circulation, and enhance joint mobility. Each paraffin wax session will last 15-20 minutes. Following the thermotherapy, participants will perform standard care exercises targeting knee mobility, flexibility, and strength. These sessions will also occur 3 times per week over a period of 8 weeks.
  Arms: Parafin Wax Bath

SUMMARY:
Knee traumas termed as any injury or damage to the knee's joint which is caused by different factors like sports injury, accidents and by fall .Knee stiffness is a common complication of femoral and tibia fracture and injuries to the extensor mechanism of the knee.

DETAILED DESCRIPTION:
There are many types of trauma of knee joint such as anterior cruciate ligament (ACL) tear, posterior cruciate ligament (PCL) tears, medial collateral ligament (MCL) tear, lateral collateral ligament (LCL) tear and meniscal tears etc. Post-traumatic knee stiffness is a commonest problem after knee injuries or surgical procedure. It affects significantly patient's quality of life and making daily living activities challenging. Paraffin wax bath therapy involves soaking targeted area in a warm paraffin wax bath pour hot liquid form wax on target area.The heat from the wax increase blood circulation in the affected areas. Mobilization with Movement (MWM) is a type manual therapy technique includes combination of joint mobilization with movement to improve joint mobility, decrease pain and improve functional ability. MWM play a role of application of joint mobilization and active movement simultaneously. The researcher employs a randomized controlled trial methodology.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years.
* Both Male and female
* Fracture of the unilateral knee joint and around the knee managed with conservative treatment only.
* Subjects with post-traumatic stiffness of knee joint having a minimum of 70º knee flexion.
* Able to walk independently or with minimal assistance.
* Administer patient in study after 12 weeks of knee injury.

Exclusion Criteria:

* deformity of hip and knee.
* Implant at fracture and around fracture site.
* Subject having polyarthritis, bleeding disorders, tumors, local infection, peripheral vascular disease, leg-length discrepancy of more than one-half inch.
* History of knee replacement or other knee surgeries within the last six months.
* Presence of neurological conditions (e.g., stroke, multiple sclerosis) affecting gait or knee mobility.
* Known allergy or intolerance to paraffin wax therapy or other study interventions."

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
VISUAL ANALOG SCALE (VAS) | 12 Months
  The Visual Analogue Scale (VAS) uses a 10 cm line with anchors like "no pain" and "worst pain imaginable", and the score is determined by measuring the distance (in mm or cm) from the "no pain" end to the patient's mark, ranging from 0 to 100
OSTEOARTHRITS INDEX (WOMAC) | 12 Months
  The Oswestry Disability Index (ODI) is a questionnaire used to assess functional disability in individuals with low back pain, with scores ranging from 0% (no disability) to 100% (maximum disability), and interpreted as follows: 0-20% minimal disability, 21-40% moderate, 41-60% severe, 61-80% crippling, and 81-100% bed-bound or exaggerated symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Shoukat ismail medical complex, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No